CLINICAL TRIAL: NCT01361919
Title: The Benefits of a Simplified Method for CPR Training of Medical Professionals: A Randomized Controlled Study
Brief Title: Three Different Cardiopulmonary Resuscitation (CPR) Training Methods
Acronym: BLSPilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: PLP 6534
Record Dates: First submitted 2010-08-03; First posted 2011-05-27 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-05

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: compressions; quality; teaching method; feedback; CPR performance; Cardiopulmonary resuscitation (CPR)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Feedback During CPR Training and Testing (Experimental): A "feedback" defibrillator (ZOLL R series) will be used at teaching, immediate testing and 12 week (retention) testing. A simulation manikin with an attached accelerometer pad on its sternum will be used to collect CPR performance data. Subjects will be told to perform compressions on top of the accelerometer pad and will be taught to use and follow the audio and visual feedback to optimize their CPR performance. After training, the raw data collected by the accelerometer will be used as a demonstration and training tool, to correct the subjects' performance by visually demonstrating the difference between ideal and suboptimal CPR performance. Testing will be carried out with the use of a "feedback" defibrillator.
  Interventions: Procedure: Feedback During CPR Training and Testing; Procedure: Feedback during CPR Training Not Testing
- Feedback during CPR Training Not Testing (Active Comparator): A "feedback" defibrillator will be used for teaching, with a standard no "feedback" defibrillator used at immediate and 12 week (retention) testing to assess if the techniques the students' learned during training are transferable to devices without "feedback". In order to collect CPR performance data, a simulation manikin with an attached accelerometer pad hidden from view within its chest will be used. Subjects will be told to perform compressions on top of the manikin's chest.
  Interventions: Procedure: Feedback During CPR Training and Testing
- No Feedback Group (Placebo Comparator): A standard no "feedback" defibrillator (ZOLL M series) will be used for teaching, immediate testing and 12 week (retention) testing. In order to collect CPR performance data, a simulation manikin with an attached accelerometer pad hidden from view within its chest will be used. Subjects will be told to perform compressions on top of the manikin's chest. During the test, subjects will be informed that data on their performance will be recorded but they will not be told how this will occur.
  Interventions: Procedure: No Feedback Group

INTERVENTIONS:
Procedure: Feedback During CPR Training and Testing — Students in this group will receive training in BLS skills according to the 2005 AHA/ILCOR guidelines, using the ZOLL R Series™ defibrillator with an attached accelerometer pad that will be placed on the sternum of the manikin and visible to the user. Participants will be taught to use and follow the audio and visual feedback provided by the accelerometer and defibrillator to optimize their CPR performance (depth, rate, and minimal "hands-off" time). After the simulated cardiac arrest scenario, a data card containing the raw data collected from the accelerometer and defibrillator will be downloaded onto a laptop and used as a demonstration and training tool.
  Arms: Feedback During CPR Training and Testing; Feedback during CPR Training Not Testing
Procedure: No Feedback Group — A standard no "feedback" defibrillator (ZOLL M series) will be used for teaching, immediate testing and 12 week (retention) testing. In order to collect CPR performance data, a simulation manikin with an attached accelerometer pad hidden from view within its chest will be used. Subjects will be told to perform compressions on top of the manikin's chest. During the test, subjects will be informed that data on their performance will be recorded but they will not be told how this will occur.
  Other Names: simulation CPR training
  Arms: No Feedback Group
Procedure: Feedback during CPR Training Not Testing — Students in this group will be tested using a five minute basic vfib arrest scenario and an R-series defibrillator and told to perform compressions on top of the accelerometer pad. The hexagonal icon will be visible but no prompting on its usage will be delivered during testing.
  Other Names: Feedback during simulation testing
  Arms: Feedback During CPR Training and Testing

SUMMARY:
The goal of this study is to compare three methods of teaching medical and nursing students basic life saving skills. The standard method will teach students how to push on the chest and to analyze the heart rhythm using a regular monitor. The newer approach will teach the same skills but use a special heart monitor that provides both visual and verbal reminders. The third approach will combine both the standard and newer approaches to teaching. Our study would like to find out the better way to teach these skills and to create a standard way to grade how well students perform. This study will measure how deep and how fast the students push on the manikin's chest in a certain amount of time. Other goals include measuring how well the students use the heart monitor to deliver shocks and analyze the heart rhythm, how many breaths per minute they give, how long their hands are off the manikin and how well they think they performed overall.

DETAILED DESCRIPTION:
The survival rates for out-of-hospital cardiac arrest (OCA) remain low (approximately 5%), despite recent advances in advanced cardiac life support (ACLS) and expansion of emergency medical services (EMS) across Ontario and Canada. Although the survival rates for in-hospital cardiac arrest are higher, less than 20% ultimately survive to discharge. One of the most important determinants of survival from cardiac arrest appears to be initiation of early and effective chest compressions. Yet the quality of cardiopulmonary resuscitation (CPR) and basic life support (BLS) delivered by first responders is often poor. CPR appears to be delivered inconsistently, incompletely and with undue delays in both the in-hospital and out-of-hospital setting. In an effort to improve cardiac arrest outcomes, focus has recently shifted to methods for training in CPR. Optimal BLS (involving chest compressions, artificial ventilation, and the use of an automated external defibrillator where available) is difficult to perform well, to teach, and to retain at a high skill level. Most BLS training programs use hands-on instruction, printed materials, and global assessment for evaluation, which to date have not been shown to impact on the quality of the CPR/BLS provided. Guidelines for BLS have changed substantially since 2005, and the efficacy of the teaching programs aimed at laypersons or primary providers of emergency care is unknown. A potential result of these limitations in the teaching, training, evaluation, and retention of BLS skills is that CPR continues to be poorly performed both by trained lay rescuers and professional caregivers.

New technologies incorporated into commercially available defibrillators may help in the training and evaluation of BLS skills. These devices allow measurement of chest compression depth and rate and ventilation frequency with continuous real-time feedback provided to the caregiver by means of an on-screen icon, which is a simple visual measure of integrated CPR efficacy, as well as verbal prompts to encourage best performance. Electronic information is stored in the defibrillator for subsequent off-line analysis which can be used to provide additional visual feedback. Perhaps most importantly, these tools provide a quantitative measure of the quality of the resuscitation effort by integrating the various aspects of CPR performance.

To date no clinical study has assessed if such tools would facilitate both the training and testing of CPR skills using the new 2005 cardiac arrest guidelines. To answer this question, the investigators propose to conduct a clinical trial involving medical and nursing students (considered "lay rescuers"), randomized to three different teaching strategies. The advantage of this population is that they are relatively easy to access and in addition, provide a homogeneous population with similarities in background, education, motivation and personal expectations. They also represent a large proportion of individuals who, in time, will be exposed to and will respond to in-hospital cardiac arrests. By using medical and nursing students who are still in the formative stages of their concepts of allied health members, the investigators hope to provide an opportunity for them to work with, about and from each other.

The control group will receive standard teaching of BLS according to the ILCOR 2005 Guidelines, including appropriate chest compression rate, depth, and chest recoil with minimization of "hands-off" time, appropriate ventilation, and use of a standard defibrillator (Zoll M series). The first intervention group will receive training supplemented by the use of a novel defibrillator (Zoll R Series) which allows for real-time continuous feedback with both visual and audio prompts to optimize CPR performance, as well as additional off-line review of details of chest compressions (including rate and depth), "hands-off" time (time spent not doing chest compressions), and therapy sequencing. The second intervention group will receive training with the novel defibrillator (Zoll R Series) but will be tested with the standard defibrillator (Zoll M series).

Two hundred and forty consenting students will be randomly assigned to the standard training ("control") group, or to training and testing using the advanced feedback features ("intervention group 1"), or to training using the advanced feedback features but tested using the standard defibrillator ("intervention group 2"), in groups of 2. After a two hour training period all participants will be tested for approximately 5 minutes. Students in the control and intervention groups will be randomized to three groups: R-Series, R series and M series or M-Series defibrillators and tested using a scenario similar to the training session.

The primary outcome is total CPR fraction (percentage of time doing chest compressions during the scenario). Secondary outcomes are CPR fraction per minute, average rate of compressions per minute, total recorded hands-off time, average depth of compressions, and the average integrated "icon fullness" as an approximation of cardiac output. Overall performance in terms of integrated psychomotor skills, reasons for hands-off time, appropriate versus inappropriate use of the AED in terms of rhythm analysis, shock delivery and study participant self-assessment of performance will also be measured. After a 3 month period, students will be re-tested using the same testing scenario to assess for skill retention. No further BLS training will be given prior to retesting.

This will be the first study to evaluate objectively and in a controlled manner the usefulness of these new technologies in the teaching, learning and evaluation of CPR/BLS.

ELIGIBILITY:
Inclusion Criteria:

* medical or nursing students aged >= 18

Exclusion Criteria:

* unwilling to sign consent, or
* unable to return in 3 months time for follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dorian, MD, FRCPC, Principal Investigator — Unity Health Toronto; Natalie Wong, MD, FRCPC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No sharing is planned

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: some participants did not record some of the baseline data elements prior to being assigned
Groups:
- Feedback During CPR Training and Testing: A "feedback" defibrillator (ZOLL R series) will be used at teaching, immediate testing and 12 week (retention) testing. A simulation manikin with an attached accelerometer pad on its sternum will be used to collect CPR performance data. Subjects will be told to perform compressions on top of the accelerometer pad and will be taught to use and follow the audio and visual feedback to optimize their CPR performance. After training, the raw data collected by the accelerometer will be used as a demonstration and training tool, to correct the subjects' performance by visually demonstrating the difference between ideal and suboptimal CPR performance. Testing will be carried out with the use of a "feedback" defibrillator.
  Feedback during CPR training: Students in this group will receive training in BLS skills according to the 2005 AHA/ILCOR guidelines, using the ZOLL R Series™ defibrillator with an attached accelerometer pad that will be placed on the sternum of the manikin and visible to
- Feedback During CPR Training Not Testing: A "feedback" defibrillator will be used for teaching, with a standard no "feedback" defibrillator used at immediate and 12 week (retention) testing to assess if the techniques the students' learned during training are transferable to devices without "feedback". In order to collect CPR performance data, a simulation manikin with an attached accelerometer pad hidden from view within its chest will be used. Subjects will be told to perform compressions on top of the manikin's chest.
  Feedback during CPR training: Students in this group will receive training in BLS skills according to the 2005 AHA/ILCOR guidelines, using the ZOLL R Series™ defibrillator with an attached accelerometer pad that will be placed on the manikin's sternum and is visible to the user. Students will be told to perform compressions on top of the accelerometer pad. Participants will be taught to use and follow the audio and visual feedback provided by the accelerometer and defibrillator to optimize their CPR perf
- No Feedback Group: A standard no "feedback" defibrillator (ZOLL M series) will be used for teaching, immediate testing and 12 week (retention) testing. In order to collect CPR performance data, a simulation manikin with an attached accelerometer pad hidden from view within its chest will be used. Subjects will be told to perform compressions on top of the manikin's chest. During the test, subjects will be informed that data on their performance will be recorded but they will not be told how this will occur.
  No Feedback during CPR Testing or Training: A standard no "feedback" defibrillator (ZOLL M series) will be used for teaching, immediate testing and 12 week (retention) testing. In order to collect CPR performance data, a simulation manikin with an attached accelerometer pad hidden from view within its chest will be used. Subjects will be told to perform compressions on top of the manikin's chest. During the test, subjects will be informed that data on their performance will be recorded.
Period: Overall Study
Arm/Group | Feedback During CPR Training and Testing | Feedback During CPR Training Not Testing | No Feedback Group
Started | 100 | 100 | 98
Completed | 90 | 88 | 88
Not Completed | 10 | 12 | 10
Not completed — technical issues | 10 | 12 | 10

BASELINE CHARACTERISTICS:
Population: All enrolled participants (n=298) completed baseline measures, however, due to technical difficulties - outcomes were not able to be collected for 32 participants as outlined above.
Groups:
- Feedback During CPR Training Not Testing: A "feedback" defibrillator will be used for teaching, with a standard no "feedback" defibrillator used at immediate and 12 week (retention) testing to assess if the techniques the students' learned during training are transferable to devices without "feedback". In order to collect CPR performance data, a simulation manikin with an attached accelerometer pad hidden from view within its chest will be used. Subjects will be told to perform compressions on top of the manikin's chest. Participants will be taught to use and follow the audio and visual feedback provided by the accelerometer and defibrillator to optimize their CPR perfor
- No Feedback Group: A standard no "feedback" defibrillator (ZOLL M series) will be used for teaching, immediate testing and 12 week (retention) testing. In order to collect CPR performance data, a simulation manikin with an attached accelerometer pad hidden from view within its chest will be used. Subjects will be told to perform compressions on top of the manikin's chest. During the test, subjects will be informed that data on their performance will be recorded but they will not be told how this will occur.
  No Feedback during CPR Testing or Training: A standard no "feedback" defibrillator (ZOLL M series) will be used for teaching, immediate testing and 12 week (retention) testing. In order to collect CPR performance data, a simulation manikin with an attached accelerometer pad hidden from view within its chest will be used. Subjects will be told to perform compressions on top of the manikin's chest.
- Total: Total of all reporting groups
Arm/Group | Feedback During CPR Training and Testing | Feedback During CPR Training Not Testing | No Feedback Group | Total
Number analyzed (Participants) | 100 | 100 | 98 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (4.1) | 24.3 (3.8) | 23.7 (3.2) | 23.8 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Some questionnaires were missing
  Participants
    number analyzed (Participants) | 98 | 99 | 98 | 295
    Female | 75 | 74 | 73 | 222
    Male | 23 | 25 | 25 | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 90 | 88 | 88 | 266
Medical Student [Count of Participants; unit: Participants] | 51 | 49 | 54 | 154
Height [Mean (Standard Deviation); unit: centimeters] | 166.8 (9.8) | 167.2 (9.8) | 167.1 (8.7) | 167.0 (9.4)
BLS Certified [Count of Participants; unit: Participants] | 89 | 86 | 91 | 266
ACLS Certified [Count of Participants; unit: Participants] | 3 | 2 | 4 | 9
Nursing Student [Count of Participants; unit: Participants] | 47 | 50 | 44 | 141

OUTCOME MEASURES:

1. Primary Outcome: CPR Depth
Description: Depth of chest compressions measured in millimeters
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Feedback During CPR Training and Testing | Feedback During CPR Training Not Testing | No Feedback Group
Number analyzed (Participants) | 90 | 88 | 88
millimeters | 43.7 (5.8) | 42.2 (6.6) | 35.3 (7.6)

2. Primary Outcome: CPR Rate
Description: rate of chest compression per minute
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: compressions per minute
Arm/Group | Feedback During CPR Training and Testing | Feedback During CPR Training Not Testing | No Feedback Group
Number analyzed (Participants) | 90 | 88 | 88
compressions per minute | 108 (7) | 105 (8) | 107 (8)

3. Secondary Outcome: Ventilations
Description: ventilations per minute over 5 minute test sequence and overall number for 5 minutes
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: number per minute
Arm/Group | Feedback During CPR Training and Testing | Feedback During CPR Training Not Testing | No Feedback Group
Number analyzed (Participants) | 90 | 88 | 88
number per minute | 20 (2) | 18 (3) | 19 (3)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Feedback During CPR Training and Testing | Feedback During CPR Training Not Testing | No Feedback Group
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/98
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/98

LIMITATIONS AND CAVEATS:
Participants' resuscitation skills were not assessed prior to providing training. The study was conducted in a simulation environment and performance in a real cardiac arrest would need to be assessed to determine the true impact of our intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No